CLINICAL TRIAL: NCT03414879
Title: Ketamine Versus Lidocaine Nebulization for Awake Nasal Fiberoptic Intubation: a Prospective, Randomized Double-blinded Study
Brief Title: Ketamine Versus Lidocaine Nebulization for Awake Fiberoptic Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Ahmad Alsayed Abdellatif, Assistant Professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R3/2018
Record Dates: First submitted 2018-01-21; First posted 2018-01-30 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ketamine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Active Comparator): Nebulization with ketamine
  Interventions: Drug: Ketamine
- Lidocaine group (Active Comparator): Nebulization with with lidocaine
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Ketamine — While in the semi-setting position, patients will receive nebulization with ketamine 3 mg/kg to be completed with normal saline solution to reach a volume of 6 ml (K group; n=30) for 15 minutes before commencing the awake fiberoptic intubation..
  Other Names: Ketalar
  Arms: Ketamine group
Drug: Lidocaine — While in the semi-setting position, patients will receive nebulization with lidocaine 4% 6 ml (L group; n=30) for 15 minutes before commencing the awake fiberoptic intubation
  Other Names: xylocaine
  Arms: Lidocaine group

SUMMARY:
This randomized double-blinded study is performed to compare ketamine versus lidocaine for nebulization for awake nasal fiberoptic intubation as regard efficacy and side effects.

DETAILED DESCRIPTION:
Difficult airway is one of the major challenges facing anesthesiologists. This challenge is compounded when the patient is treated while awake. The additional burden is to complete this procedure comfortably thus ensuring patient cooperation which is a vital part of successful performance. Several methods have been tried in literature to facilitate awake intubation by fiberoptic bronchoscope (FOB)

This randomized double-blinded study is performed to compare ketamine versus lidocaine for nebulization for awake nasal fiberoptic intubation as regard efficacy and side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I and II of both sexes with body weight from 60-90 kg, and planned for elective awake nasal fiberoptic intubation due to expected difficulty in airway management (e.g. limited mouth opening, trismus, mandibular/ maxillary swellings or tumors, ludwig's angina, or other indications).

Exclusion Criteria:

* body weight < 60 kg or > 90 kg
* uncooperative, with mental or psychological problems
* known allergy to any of the study drugs
* pregnancy
* hypertension
* cardiac disease
* liver or renal impairment
* epilepsy,
* asthmatic,
* previous bad experience of awake intubation,
* emergency operations or
* coagulation abnormalities

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Dose of supplemental lidocaine | Intraoperative
  Dose of supplemental lidocaine during awake fiberoptic procedure

SECONDARY OUTCOMES:
Incidence of adverse events | Intraoperative
  The incidence of adverse events related to the procedure and study drugs will be recorded
Patient satisfaction score | first 24 hours
  will be assessed against five point Likert score where (1: poor, 2: fair, 3: good, 4: very good, 5: excellent).
Patient tolerability score | Intraoperative
  Patient tolerability during the procedure will be rated as 4-point scale where 0= procedure totally intolerable with severe patient resistance (struggling/withdrawal movements).
  1. procedure partially tolerable with moderate patient resistance (restlessness/ verbal objection).
  2. procedure quiet tolerable with minimal patient resistance (just grimacing).
  3. procedure tolerable with no patient resistance. this score will be recorded at points during the intubation procedure: nasal passage, oro/hypopharynx, glottis and tube insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No